CLINICAL TRIAL: NCT00834899
Title: A Phase I/II Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety of Eptifibatide as Treatment for Acute Pain Episodes in Sickle Cell Disease
Brief Title: A Safety Study of Eptifibatide in Patients With Sickle Cell Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual and no cost extension not approved by NHLBI
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R21HL091265-01A1 (NIH)
Record Dates: First submitted 2009-01-31; First posted 2009-02-03 (Estimated); Results first posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-02

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Pain crisis; Acute pain episode; Eptifibatide; Antiplatelet therapy; Safety; Treatment
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Eptifibatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): As soon as eligible patients are identified and provide consent to participate in the study, patients randomized to the eptifibatide arm will receive two 180 mcg/kg boluses of eptifibatide 10 minutes apart (i.e., a double bolus), followed by a continuous infusion at 2 mcg/kg/min for 6 hours.
  Interventions: Drug: Eptifibatide
- 2 (Placebo Comparator): As soon as eligible patients are identified and provide consent to participate in the study, patients randomized to the placebo arm will receive a saline solution delivered at a volume and rate identical to that of the active drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eptifibatide — Patients randomized to eptifibatide will receive two 180 mcg/kg boluses of eptifibatide 10 minutes apart (i.e., a double bolus), followed by a continuous infusion at 2 mcg/kg/min for 6 hours.
  Other Names: Integrilin
  Arms: 1
Drug: Placebo — Patients randomized to the placebo arm will receive a saline solution delivered at a volume and rate identical to that of the active drug.
  Arms: 2

SUMMARY:
This study will evaluate the safety of eptifibatide in sickle cell patients and how well it works during the course of painful crises. The overall hypothesis that we seek to test is that increased platelet activation and the resultant inflammatory responses are important contributors to the problems of sickle cell disease. Sickle cell disease has been referred to both as a condition associated with increased risk of blood clots and increased inflammation. A painful crisis represents the most common cli nical problem in sickle cell disease, but the treatment of these crises remains inadequate.

DETAILED DESCRIPTION:
Sickle cell disease has been referred to both as a condition associated with increased risk of blood clots and increased inflammation. Despite the abundant laboratory evidence of abnormal blood clotting and inflammation, the contribution of these changes to the problems experienced by patients with sickle cell disease remains uncertain. In additional to abnormal blood clotting, platelets (small blood cells that help blood clotting) are more activated in sickle cell disease patients compared to healthy patients without this disease.

In addition, when sickle cell disease patients experience a painful crisis, there is evidence that the platelet activation and abnormal blood clotting increase even further. Activated platelets release a substance called cluster of designation 40 ligand, which can increase how sticky the lining of blood vessels are and can increase the abnormal blood clotting. The level of cluster of designation 40 ligand is much higher in sickle cell disease patients compared to healthy individuals without this disease. In addition, the levels increase even further when sickle cell patients are experiencing a painful crisis.

Painful crisis represent the most common clinical problem in sickle cell disease, and are largely responsible for making the lives of these patients so unpredictable. However, the treatment of these painful crisis remains inadequate, consisting mainly of strong pain medications. In this study, we will evaluate the safety of eptifibatide in sickle cell patients and how well it works during the course of painful crises. At the completion of this trial, we will have an improved understanding of the contribution of platelet activation and inflammation to the problems in sickle cell disease.

The overall hypothesis that we seek to test is that increased platelet activation and the resultant inflammatory responses are important contributors to the problems of sickle cell disease. We believe that by decreasing platelet stickiness, and the release of mediators of inflammation and abnormal blood clotting, eptifibatide will affect the clinical course of complications in this disease.

If the results from our study support the hypothesis that eptifibatide is safe and effective in this population, we plan on carrying out larger studies to more definitively evaluate the safety of eptifibatide and how well it works in the treatment and/or prevention of painful crises in sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 55 years
2. Have confirmed diagnosis of sickle cell anemia or sickle beta zero thalassemia
3. Have a serum creatinine </= 1.2 mg/dl
4. Have serum transaminase values < 3 times upper limits of normal
5. Have a platelet count >/= 150 x 10^9/L
6. Have normal baseline coagulation profile
7. Sudden onset of pain involving one or more sites and typical of usual pain episodes
8. Have adequate intravenous access
9. Be able to understand the requirements of the study and be willing to give informed consent
10. Women of child-bearing age must be practicing (and will continue to practice for the course of the study) an adequate method of contraception (oral contraception, depo-provera, bilateral tubal ligation or barrier method)

Exclusion Criteria:

1. Have a baseline hemoglobin < 6.0 gm/dl
2. Have a history of major gastrointestinal bleeding or a bleeding diathesis
3. Have an ongoing episode of acute chest syndrome
4. Have a past history of clinically overt stroke(s)
5. Have severe hypertension (systolic blood pressure > 200mmHg and/or diastolic BP >110mmHg) not adequately controlled on hypertensive medication
6. Have had major surgery within the six weeks preceding enrollment
7. Are pregnant or breastfeeding
8. Are on chronic anticoagulation or antiplatelet (including non-steroidal anti-inflammatory drugs) therapy
9. Have a history of metastatic cancer
10. Are on a chronic transfusion program or have received a blood transfusion in the prior 8 weeks
11. Have a positive urine toxicology screen for phencyclidine, cocaine or amphetamines.
12. Have a history of alcohol abuse
13. Have received any investigational drugs within the past 4 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth I Ataga, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Desai PC, Brittain JE, Jones SK, McDonald A, Wilson DR, Dominik R, Key NS, Parise LV, Ataga KI. A pilot study of eptifibatide for treatment of acute pain episodes in sickle cell disease. Thromb Res. 2013 Sep;132(3):341-5. doi: 10.1016/j.thromres.2013.08.002. Epub 2013 Aug 8. PMID 23973010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with sickle cell disease, admitted with an acute pain episode, and who met eligibility criteria were approached to participate.
Pre-assignment Details: Patient who agreed to participate provided informed consent and were screened for eligibility. Eligible patients were subsequently randomized to treatment with eptifibatide or placebo.
Groups:
- Eptifibatide: Patients randomized to the eptifibatide arm received two 180 mcg/kg boluses of eptifibatide 10 minutes apart (i.e., a double bolus), followed by a continuous infusion at 2 mcg/kg/min for 6 hours.
- Placebo: Patients randomized to the placebo arm received a saline solution delivered at a volume and rate identical to that of the active drug.
Period: Overall Study
Arm/Group | Eptifibatide | Placebo
Started | 9 | 4
Completed | 8 (One patient withdrew consent following completion of the study drug infusion.) | 3 (One patient was withdrawn early because she did not meet eligibility criteria.)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eptifibatide | Placebo | Total
Number analyzed (Participants) | 9 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 4 | 13
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.6 (8.78) | 34.0 (12.19) | 31.6 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 4 | 13
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: 1) Major Bleeding Episodes
Description: Major bleeding episodes are defined as any episode, such as gastrointestinal bleeding or intracranial bleed that typically leads to hospitalization or other prolonged bleeding requiring a blood transfusion
Time Frame: Up to 35 days
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Eptifibatide | Placebo
Number analyzed (Participants) | 9 | 4
participants | 0 [-0.604 to 0.372] | 0 [-0.604 to 0.372]

2. Secondary Outcome: Effect of Eptifibatide on Duration of Acute Pain Episodes
Description: The duration of the pain episode will be defined as the time from randomization to termination of the pain episode. The pain episode will be considered terminated when the patient states that the crisis is resolved (defined as being ready to go home on oral analgesics) or all of the following criteria are met:
  1. Pain relief (pain scores ≤ 40) maintained for at least 2 consecutive readings (assessed using a visual analog scale with measurements from 0 - 100, where 0 is no pain and 100 is worst imaginable pain).
  2. No parenteral analgesics have been administered for at least 12 hours.
  3. Ability to walk normally (unless he/she was unable to walk for some other reason prior to the crisis onset).
Time Frame: Up to 7 days
Population: Intention to treat
Measure: Median (Full Range); unit: Days
Arm/Group | Eptifibatide | Placebo
Number analyzed (Participants) | 9 | 4
Days | 3.0 [1.81 to 8.0] | 3.0 [0.08 to 3.92]

3. Secondary Outcome: Effect of Eptifibatide on Duration of Hospitalization
Description: The duration of hospitalization will be defined as the period from randomization to the time an order for discharge from the hospital is written.
Time Frame: Up to 7 days
Population: Intention to treat
Measure: Median (Full Range); unit: Days
Arm/Group | Eptifibatide | Placebo
Number analyzed (Participants) | 9 | 4
Days | 3.0 [2.0 to 36.1] | 3.0 [2.0 to 4.0]

4. Primary Outcome: Change in Platelet Count
Description: Change in platelet counts occurring anytime from randomization up to day 35 (final follow-up visit).
Time Frame: Up to 35 days
Measure: Median (Full Range); unit: x 10^9/L
Arm/Group | Eptifibatide | Placebo
Number analyzed (Participants) | 9 | 4
x 10^9/L | 97 [-50 to 410] | -5 [-63 to 129]

ADVERSE EVENTS:
Arm/Group | Eptifibatide | Placebo
Serious Adverse Events (participants affected / at risk) | 8/9 | 2/4
Other Adverse Events (participants affected / at risk) | 7/9 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptifibatide (N=9) | Placebo (N=4)
Adenovirus Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bacteremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypoxemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Shoulder Pain, Left (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder Pain, Right (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sickle Cell Crisis, recurrent (Blood and lymphatic system disorders) | 3 (4) | 1 (1)
Worsening anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Chest Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptifibatide (N=9) | Placebo (N=4)
Ankle Swelling, bilateral (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Excessive perspiration (General disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 2 (3)
Headache, recurrent (Nervous system disorders) | 1 (1) | 0 (0)
Infusion site extravasation (Vascular disorders) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nosebleed (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Possible Acute Chest Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Reticulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sickle Cell Crisis, recurrent (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Sickle Cell Crisis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sore Throat (General disorders) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early resulting in small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No